CLINICAL TRIAL: NCT04243551
Title: Multicenter, Prospective, Randomized, Double-Blind, Placebo-Controlled, Crossover Study of the Efficacy and Safety of Latiglutenase Treatment in Symptomatic Celiac Disease Patients Maintained on a Gluten-Free Diet While Undergoing Periodic Gluten Exposure
Brief Title: Prospective, Randomized, Double-Blind, Placebo-Controlled, Crossover Study in Symptomatic CD Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to low enrollment related to Covid.
Sponsor: Entero Therapeutics (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IMGX003-NIAID-1821; U44AI134590 (NIH)
Record Dates: First submitted 2020-01-23; First posted 2020-01-28 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2023-07

CONDITIONS: Celiac Disease
Keywords: Celiac
MeSH Terms: conditions — Celiac Disease | interventions — ALV003

STUDY DESIGN:
Intervention Model Description: A two-period crossover design will be used where the two possible treatment sequences will be assigned at random.
Who Masked: Participant, Investigator
Masking Description: The PI, CRA and study biostatistician will be masked until database lock.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Latiglutenase (Active Comparator): IMGX003
  Interventions: Drug: Latiglutenase
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Latiglutenase — Administered orally (daily)
  Other Names: IMGX003
  Arms: Latiglutenase
Other: Placebo — Administered orally (daily)
  Arms: Placebo

SUMMARY:
This is a phase 2b, multicenter, prospective, randomized, double-blind, placebo-controlled, crossover study in symptomatic celiac disease patients attempting a GFD for at least one year prior to screening.

DETAILED DESCRIPTION:
This is a phase 2b, multicenter, prospective, randomized, double-blind, placebo-controlled, crossover study in symptomatic celiac disease patients attempting a GFD for at least one year prior to screening. Seropositive patients (blood test confirmed at Visit 0) will be scheduled for a Screening Visit (Visit 1) whereas seronegative patients will be discontinued from study participation (screen failures). Patients who meet Visit 1 protocol enrollment criteria will be enrolled and begin the first of two 6 week periods.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy confirmed CD diagnosis
* Seropositive
* Gluten free diet (12 months minimum)
* Experienced at least one self reported moderate or greater severity symptom during the last 28 day period
* Willing to take study treatment daily
* Must sign informed consent

Exclusion Criteria:

* Wheat allergy
* History of peptic ulcer disease, esophagitis, IBS, IBD
* Active colitis, dermatitis herpetiformis
* Diagnosed with Type 1 Diabetes
* Patients with known rapid gastric emptying (post-bariatric surgery, Billroth I or II surgery)
* Chronic infectious gastrointestinal illness or acute infectious gastrointestinal illness within the 4 week period prior to screening
* Known refractory celiac disease (RCD1 or RCD2)
* Inability to give informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2023-10-16 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Symptom Severity Reduction | 6 months
  The primary efficacy endpoint of this study is mean percent reduction in symptom severity relative to placebo.

SECONDARY OUTCOMES:
Health Related Quality of Life | 6 months
  A secondary efficacy endpoint includes a change from baseline to end of study treatment period in health-related quality of life as measured by PGI-I health survey relative to placebo.
Health Related Quality of Life | 6 months
  A secondary efficacy endpoint includes a change from baseline to end of study treatment period in health-related quality of life as measured by PGI-S health survey relative to placebo.
Health Related Quality of Life | 6 months
  A secondary efficacy endpoint includes a change from baseline to end of study treatment period in health-related quality of life as measured by ICDSQ health survey relative to placebo.
Health Related Quality of Life | 6 months
  A secondary efficacy endpoint includes a change from baseline to end of study treatment period in health-related quality of life as measured by SF-12 health survey relative to placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Murray, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No